CLINICAL TRIAL: NCT07011511
Title: A First-in-Human, Single-Centre, Single Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of Intramuscular Injection(s) of Long-Acting Injectable Formulations of MMV055 Alone (Part A) and in Combination With MMV371 (Part B) in Healthy Participants
Brief Title: Single Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of LAI MMV055 Alone and in Combination With MMV371 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Quotient Sciences (Industry); The Doctors Laboratory Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: MMV_MMV055_24_01_FIH
Record Dates: First submitted 2025-05-19; First posted 2025-06-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Malaria, Falciparum
Keywords: Malaria; First In Human; Healthy Volunteers
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part A1 Regimen A (Experimental)
  Interventions: Drug: MMV055 Dose 1; Drug: Matching placebo Part A
- Part A1 Regimen B (Experimental)
  Interventions: Drug: MMV055 Dose 2; Drug: Matching placebo Part A
- Part A2 Regimen C (Experimental)
  Interventions: Drug: MMV055 Dose 3; Drug: Matching placebo Part A
- Part A2 Regimen D (Experimental)
  Interventions: Drug: MMV055 Dose 4; Drug: Matching placebo Part A
- Part A2 Regimen E (Experimental)
  Interventions: Drug: MMV055 Dose 5; Drug: Matching placebo Part A
- Part A2 Regimen F (Experimental)
  Interventions: Drug: MMV055 Dose 6; Drug: Matching placebo Part A
- Part B Combination 1 (Experimental)
  Interventions: Drug: Matching placebo Part B; Combination Product: MMV055/MMV371 Combo 1
- Part B Combination 2 (Experimental)
  Interventions: Drug: Matching placebo Part B; Combination Product: MMV055/MM371 Combo 2
- Part B Combination 3 (Experimental)
  Interventions: Drug: Matching placebo Part B; Combination Product: MMV055/MMV371 Combo 3

INTERVENTIONS:
Drug: MMV055 Dose 1 — 40mg
  Arms: Part A1 Regimen A
Drug: MMV055 Dose 2 — 100mg
  Arms: Part A1 Regimen B
Drug: MMV055 Dose 3 — 200mg
  Arms: Part A2 Regimen C
Drug: MMV055 Dose 4 — 400mg
  Arms: Part A2 Regimen D
Drug: MMV055 Dose 5 — 800mg
  Arms: Part A2 Regimen E
Drug: MMV055 Dose 6 — TBCmg
  Arms: Part A2 Regimen F
Drug: Matching placebo Part A — Part A
  Arms: Part A1 Regimen A; Part A1 Regimen B; Part A2 Regimen C; Part A2 Regimen D; Part A2 Regimen E; Part A2 Regimen F
Drug: Matching placebo Part B — Part B
  Arms: Part B Combination 1; Part B Combination 2; Part B Combination 3
Combination Product: MMV055/MMV371 Combo 1 — Combination 1
  Arms: Part B Combination 1
Combination Product: MMV055/MM371 Combo 2 — Combination 2
  Arms: Part B Combination 2
Combination Product: MMV055/MMV371 Combo 3 — Combination 3
  Arms: Part B Combination 3

SUMMARY:
This is a single-centre, participant- and investigator-blind, randomised, placebo controlled, single ascending dose study to assess the safety, tolerability and PK of a single dose of IM depot injection(s) of LAI formulations of MMV055 administered alone (Part A) and in combination with MMV371 (Part B) in healthy participants.

It is planned to enroll up to 6 sequential cohorts of 8 healthy male participants and healthy female participants of non-childbearing potential in Part A. In Part B, up to 3 sequential cohorts of 8 healthy male participants and healthy non-pregnant, non-lactating female participants will be enrolled. In each cohort, participants will be randomised in a ratio of 6 active investigational medicinal product (IMP) to 2 placebo.

Part A of the study will include two components, Parts A1 and A2. Part A1 includes two initial cohorts, with planned doses of 40 and 100mg, respectively. It is intended to document the human elimination T1/2 of MMV055, which will then be used to shorten the proposed End of Study (EOS) of 48 weeks, if possible.

All cohorts will follow a sentinel dosing design. On Day 1, two sentinel participants (sentinel group) will be randomly assigned to receive a single IM dose of either active IMP or placebo (1 participant each) to assess safety and tolerability (including ISRs).

The sentinel group will be dosed concomitantly at least 7 days prior to the rest of the cohort (main group). The main group will comprise 6 participants randomly assigned to receive a single IM dose of either active IMP or placebo in a 5:1 ratio to assess safety and tolerability (including ISRs).

ELIGIBILITY:
Inclusion Criteria:

1. Must provide written informed consent
2. Must be willing and able to communicate and participate in the whole study
3. Aged 18 to 60 years inclusive at the time of signing informed consent
4. Must agree to adhere to the contraception requirements defined in the study protocol
5. Healthy male or healthy WONCBP (Parts A and B), or healthy non-pregnant, non-lactating female participants (Part B only) according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs, 12-lead ECG, and laboratory safety tests without any clinically significant abnormalities. Safety bloods, urinalysis, ECGs and vital signs to be re-checked at admission and/or pre-dose
6. Body mass index (BMI) of 19.0 to 30.0 kg/m2 as measured at screening
7. Weight ≥50 kg for males and ≥45 kg for females at screening

Exclusion Criteria:

1. Serious adverse reaction or serious hypersensitivity to any drug or formulation excipients (Parts A and B), Wellvone®/Mepron® and/or Malarone® (Part B only)
2. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
3. History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or GI disease, neurological or psychiatric disorder, as judged by the investigator
4. Family history of sudden death, or family history of clinically significant cardiovascular disease, as judged by the investigator
5. Systolic BP >140 or <90 mmHg, diastolic BP >90 or <50 mmHg, or heart rate (HR) (based on vital signs assessment) >100 or <45 bpm, confirmed by repeat assessment at screening
6. Any finding in the medical examination (including BP, HR or ECG) deviating from normal and assessed as clinically relevant by the investigator
7. History or presence of known structural cardiac abnormalities, family history of long QT syndrome, cardiac syncope or recurrent, idiopathic syncope, exercise related clinically significant cardiac events. Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG or clinically important abnormalities that may interfere with the interpretation of QT changes
8. Presence of sinus node dysfunction, clinically significant PR interval prolongation (>220 msec), intermittent second- or third-degree atrioventricular block, complete bundle branch block, sustained cardiac arrhythmias including (but not limited to) atrial fibrillation or supraventricular tachycardia; any symptomatic arrhythmia with the exception of isolated extra systoles, abnormal T wave morphology which may impact on the QT/QTc assessment, or QTcF >450 msec based on the mean of the triplicate values and confirmed by single repeat assessment at screening
9. Participants with a history of cholecystectomy or gall stones
10. Participants who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
11. Participants with tattoos or scars or other significant dermatological conditions overlying the deltoid or gluteal region which may interfere with injection site assessments, as determined by the investigator or delegate at screening
12. Clinically significant abnormal clinical chemistry, haematology, coagulation or urinalysis as judged by the investigator (laboratory parameters are listed in the study protocol). Participants with Gilbert's Syndrome are not allowed
13. Dyslipidaemia (cholesterol and/or triglycerides) requiring pharmacological intervention or fasting triglycerides >2.26 mmol/L, fasting cholesterol >6.20 mmol/L, low density lipoprotein cholesterol >3.75 mmol/L)
14. Fasting blood glucose ≥6.1 mmol/L
15. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) 1 and 2 antibody results
16. Transaminases (ALT or AST) >ULN
17. Females who are pregnant or lactating (all female participants must have a negative highly sensitive serum pregnancy test at screening and a negative urine pregnancy test at admission)
18. Part A only: females of childbearing potential. A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) or is post-menopausal (had no menses for 12 months without an alternative medical cause and a serum follicle stimulating hormone [FSH] concentration ≥40 IU/L).
19. Participants who have received any IMP in a clinical research study within the 90 days prior to Day 1, or less than 5 elimination half-lives prior to Day 1, whichever is longer
20. Participants who have previously been administered MMV055 in this study
21. Participants who report to have previously received MMV371
22. Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood
23. Participants who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day, up to 800 mg ibuprofen per day, hormonal contraception or HRT) in the 14 days before IMP administration (see study protocol). Exceptions may apply, as determined by the investigator, if each of the following criteria are met: medication with a short half-life if the washout is such that no pharmacodynamic activity is expected by the time of dosing with IMP; and if the use of medication does not jeopardise the safety of the trial participant; and if the use of medication is not considered to interfere with the objectives of the study.
24. Participants who are taking, or who have taken, rifampin/rifabutin, tetracycline and indinavir in the 30 days before IMP administration (Part B only)
25. Live vaccines within 30 days of IMP administration, or plans to receive such vaccines during the study
26. Participants who have had a COVID 19 vaccine within 14 days before dosing
27. History of any drug or alcohol abuse in the past 2 years
28. Regular alcohol consumption in males >21 units per week and in females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type)
29. A confirmed positive alcohol breath test at screening or admission
30. Current smokers and those who have smoked within the last 12 months
31. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
32. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
33. Confirmed positive drugs of abuse test result (drugs of abuse tests are listed in the study protocol) at screening or admission
34. Male participants with pregnant or lactating partners
35. A score of SI 4 to 5 (related to suicidal ideation) or any SB score (related to suicidal behaviour) as assessed using the Columbia-Suicide Severity Rating Scale (C SSRS)
36. Participants who are, or are immediate family members of, a study site or sponsor employee
37. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-12-02 (Estimated); Study Completion 2027-12-02 (Estimated)

PRIMARY OUTCOMES:
Safety - Incidence of AEs | From enrollment to the last follow up visit at week 56
  Number of participants with AEs
Safety - Incidence of Injection Site Reactions | From enrollment to the last follow up visit at week 56
  Number of participants with Injection Site Reactions
Safety - Incidence of physical examination findings | From enrollment to the last follow up visit at week 56
  Number of participants with physical examination findings
Safety - Vital signs changes from baseline | From enrollment to the last follow up visit at week 56
  Number of participants with clinically significant vital signs changes from baseline
Safety - ECG changes from baseline, QT intervals | From enrollment to the last follow up visit at week 56
  Number and percentage of participants with normal and prolonged QT intervals corrected for Fridericia's correction (i.e. QTcF) and increases in QTcF intervals from baseline
Safety - ECG changes from baseline, PR and QRS intervals | From enrollment to the last follow up visit at week 56
  Number and percentage of participants with clinically significant changes in PR and QRS intervals
Part 1 only: plasma concentrations of MMV055: Cmax | From enrollment to the last follow up visit at week 56
  Expressed in ng/mL
Part 1 only: plasma concentrations of MMV055: AUC(0-last) | From enrollment to the last follow up visit at week 56
  Expressed in ng.h/mL
Part 1 only: plasma concentrations of MMV055: AUC(0-inf) | From enrollment to the last follow up visit at week 56
  Expressed in ng.h/mL
Part 1 only: plasma concentrations of MMV055: T1/2 | From enrollment to the last follow up visit at week 56
  Expressed in hours

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.quotientsciences.com/volunteers